CLINICAL TRIAL: NCT04997291
Title: Use of the Cardioprotectant Dexrazoxane During Congenital Heart Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: Dell Children's Medical Center of Central Texas (Other)
Responsible Party: Principal Investigator, Daniel Stromberg, Associate Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02-0075
Record Dates: First submitted 2021-07-21; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Dexrazoxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexrazoxane (Experimental)
  Interventions: Drug: Dexrazoxane

INTERVENTIONS:
Drug: Dexrazoxane — Twelve enrollees will be consecutively assigned to a dosing regimen of 400 mg/m2/dose. The medication will be administered in the operating room 30 minutes prior to starting cardiopulmonary bypass (dose #1), prior to aortic cross clamp removal (dose #2), and on the morning after surgery in the cardiac intensive care unit (dose #3).
  Other Names: Zinecard

SUMMARY:
Cardiopulmonary bypass and arrest of the heart during cardiac surgery are necessary to allow the surgeon to perform heart operations. However, these processes can cause injury to the heart which may worsen post-operative outcomes. In fact, the effects of these injuries may continue after surgery, and lead to a long-term decrease in heart function. Neonates and young infants are at particular risk for this occurrence.

While much research has been done in adults looking for medicines that might protect the heart during surgery, few studies have been conducted in neonates and young infants. The investigators are testing Dexrazoxane, which has proven to be cardio-protective in pediatric cancer patients, in the hope that it may lessen cardiac injury during and after congenital heart surgery, and thereby improve outcomes in the neonatal and young infant population.

In order to accomplish this, the investigators must first determine how Dexrazoxane can be safely administered to young children with congenital heart disease.

DETAILED DESCRIPTION:
Neonates and infants undergoing heart surgery with cardiopulmonary bypass and cardioplegic arrest experience both inflammation and myocardial ischemia-reperfusion [IR] injury. These processes provoke myocardial apoptosis and oxygen free radical formation which result in cardiac injury and dysfunction. Dexrazoxane [DRZ] is a derivative of EDTA that is approved for prevention of anthracycline-related cardiotoxicity. It provides cardioprotection through reduction of toxic reactive oxygen species [ROS], and suppression of apoptosis.

The investigators propose a 12-patient pilot to determine DRZ pharmacokinetics, and to collect additional safety data in the neonatal and infant population. Efficacy of cardioprotection will not be evaluated in this preliminary investigation, though the investigators will determine postoperative time to resolution of organ failure, development of low cardiac output syndrome, length of cardiac ICU and hospital stays, laboratory indices of myocardial injury and systemic inflammation, and echocardiographic cardiac dysfunction for safety purposes, and as a run-in to the larger, randomized, placebo controlled trial. Conducting this pilot could optimize team execution of the study protocol. In addition, results could further establish the safety of DRZ in the neonatal and infant populations.

ELIGIBILITY:
Inclusion Criteria:

* age ≤ 1 year
* open heart surgery requiring CPB and use of cardioplegia
* parent/guardian consent for study obtained
* surgery planned Monday-Friday

Exclusion Criteria:

* gestational age <36 weeks at time of enrollment
* known syndrome or genetic abnormality, except Trisomy 21
* single ventricle physiology
* concurrent enrollment in another research protocol

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 24 hours
Area under the plasma concentration vs time curve (AUC) | 24 hours
Minimum plasma concentration (Cmin) | 24 hours
Time to resolution of organ failure | 14 days
  defined as hours to the point of being off invasive mechanical ventilation, without significant renal dysfunction [cystatin C within normal range for age, and UOP > 1 cc/kg/hr], and off significant inotropic support [defined as milrinone >0.3 mcg/kg/min, dopamine >3 mcg/kg/min, dobutamine >3 mcg/kg/min, any combination of these inotropes, or any epinephrine, norepinephrine, phenylephrine or vasopressin)] with a serum lactate <2 mmol/L. One point will be awarded for each postoperative hour of continued organ dysfunction up to postoperative hour 336 (day 14). A score of 360 will be assigned if organ failure is not resolved by postoperative day 14, or if the patient requires mechanical circulatory support or experiences mortality. This variable has been chosen to allow for recognition of early drug effects, and those which might be delayed beyond the immediate postoperative period.

SECONDARY OUTCOMES:
Myocardial Injury | 7 days
  determined by elevated serum cardiac troponin
Oxidative Stress | 3 days
  measured by lipoperoxidation (serum F2 isoprostane)
Inflammatory activation (IL-6 and IL-10) | 3 days
Neurologic IR injury | 3 days
  measured by serum activin A concentration
ICU Length of Stay | 60 days
Hospital Length of Stay | 60 days
Tei Index (via echocardiogram) | 60 days
  the sum of the isovolumic contraction and relaxation times divided by the ejection time
Ventricular ejection fraction (via echocardiogram) | 60 days
  the volumetric fraction of fluid ejected from a chamber with each contraction
Tissue doppler E/E' ratio (via echocardiogram) | 60 days
  calculated as E wave divided by e' velocities
Composite outcome for neonatal cardiac surgery | 60 days
  (per Graham, EM, et al) - binary variable defined as death, use of mechanical circulatory support, cardiac arrest requiring chest compressions, hepatic injury [2 times the upper limit of normal for AST or ALT], renal injury [Cr >1.5 mg/dL], or lactic acidosis [an increasing lactate >5 mmol/L in the postoperative period]

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Children's Medical Center of Central Texas, Austin, Texas, United States

REFERENCES:
- [Background] Chaney MA. Corticosteroids and cardiopulmonary bypass : a review of clinical investigations. Chest. 2002 Mar;121(3):921-31. doi: 10.1378/chest.121.3.921. PMID 11888978
- [Background] Caputo M, Mokhtari A, Rogers CA, Panayiotou N, Chen Q, Ghorbel MT, Angelini GD, Parry AJ. The effects of normoxic versus hyperoxic cardiopulmonary bypass on oxidative stress and inflammatory response in cyanotic pediatric patients undergoing open cardiac surgery: a randomized controlled trial. J Thorac Cardiovasc Surg. 2009 Jul;138(1):206-14. doi: 10.1016/j.jtcvs.2008.12.028. Epub 2009 Feb 23. PMID 19577081
- [Background] Hare JM. Oxidative stress and apoptosis in heart failure progression. Circ Res. 2001 Aug 3;89(3):198-200. No abstract available. PMID 11485969
- [Background] Pasquali SK, Hall M, Li JS, Peterson ED, Jaggers J, Lodge AJ, Marino BS, Goodman DM, Shah SS. Corticosteroids and outcome in children undergoing congenital heart surgery: analysis of the Pediatric Health Information Systems database. Circulation. 2010 Nov 23;122(21):2123-30. doi: 10.1161/CIRCULATIONAHA.110.948737. Epub 2010 Nov 8. PMID 21060075
- [Background] Robertson-Malt S, Afrane B, El Barbary M. Prophylactic steroids for pediatric open heart surgery. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD005550. doi: 10.1002/14651858.CD005550.pub2. PMID 17943866
- [Background] Graham EM, Atz AM, Butts RJ, Baker NL, Zyblewski SC, Deardorff RL, DeSantis SM, Reeves ST, Bradley SM, Spinale FG. Standardized preoperative corticosteroid treatment in neonates undergoing cardiac surgery: results from a randomized trial. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1523-9. doi: 10.1016/j.jtcvs.2011.04.019. Epub 2011 May 20. PMID 21600592
- [Background] Schroeder VA, Pearl JM, Schwartz SM, Shanley TP, Manning PB, Nelson DP. Combined steroid treatment for congenital heart surgery improves oxygen delivery and reduces postbypass inflammatory mediator expression. Circulation. 2003 Jun 10;107(22):2823-8. doi: 10.1161/01.CIR.0000070955.55636.25. Epub 2003 May 19. PMID 12756159
- [Background] Checchia PA, Backer CL, Bronicki RA, Baden HP, Crawford SE, Green TP, Mavroudis C. Dexamethasone reduces postoperative troponin levels in children undergoing cardiopulmonary bypass. Crit Care Med. 2003 Jun;31(6):1742-5. doi: 10.1097/01.CCM.0000063443.32874.60. PMID 12794414
- [Background] Clarizia NA, Manlhiot C, Schwartz SM, Sivarajan VB, Maratta R, Holtby HM, Gruenwald CE, Caldarone CA, Van Arsdell GS, McCrindle BW. Improved outcomes associated with intraoperative steroid use in high-risk pediatric cardiac surgery. Ann Thorac Surg. 2011 Apr;91(4):1222-7. doi: 10.1016/j.athoracsur.2010.11.005. PMID 21440149
- [Background] Clancy RR, McGaurn SA, Goin JE, Hirtz DG, Norwood WI, Gaynor JW, Jacobs ML, Wernovsky G, Mahle WT, Murphy JD, Nicolson SC, Steven JM, Spray TL. Allopurinol neurocardiac protection trial in infants undergoing heart surgery using deep hypothermic circulatory arrest. Pediatrics. 2001 Jul;108(1):61-70. doi: 10.1542/peds.108.1.61. PMID 11433055
- [Background] Jin Z, Duan W, Chen M, Yu S, Zhang H, Feng G, Xiong L, Yi D. The myocardial protective effects of adenosine pretreatment in children undergoing cardiac surgery: a randomized controlled clinical trial. Eur J Cardiothorac Surg. 2011 May;39(5):e90-6. doi: 10.1016/j.ejcts.2010.12.052. Epub 2011 Feb 20. PMID 21342773
- [Background] Walavalkar V, Evers E, Pujar S, Viralam K, Maiya S, Frerich S, John C, Rao S, Reddy C, Spronck B, Prinzen FW, Delhaas T, Vanagt WY. Preoperative Sildenafil administration in children undergoing cardiac surgery: a randomized controlled preconditioning study. Eur J Cardiothorac Surg. 2016 May;49(5):1403-10. doi: 10.1093/ejcts/ezv353. Epub 2015 Oct 13. PMID 26464453
- [Background] Wu Q, Wang T, Chen S, Zhou Q, Li H, Hu N, Feng Y, Dong N, Yao S, Xia Z. Cardiac protective effects of remote ischaemic preconditioning in children undergoing tetralogy of fallot repair surgery: a randomized controlled trial. Eur Heart J. 2018 Mar 21;39(12):1028-1037. doi: 10.1093/eurheartj/ehx030. PMID 28329231
- [Background] Tie HT, Luo MZ, Li ZH, Wang Q, Wu QC, Li Q, Zhang M. Remote Ischemic Preconditioning Fails to Benefit Pediatric Patients Undergoing Congenital Cardiac Surgery: A Meta-Analysis of Randomized Controlled Trials. Medicine (Baltimore). 2015 Oct;94(43):e1895. doi: 10.1097/MD.0000000000001895. PMID 26512608
- [Background] James C, Millar J, Horton S, Brizard C, Molesworth C, Butt W. Nitric oxide administration during paediatric cardiopulmonary bypass: a randomised controlled trial. Intensive Care Med. 2016 Nov;42(11):1744-1752. doi: 10.1007/s00134-016-4420-6. Epub 2016 Sep 30. PMID 27686343
- [Background] Ferreira R, Burgos M, Milei J, Llesuy S, Molteni L, Hourquebie H, Boveris A. Effect of supplementing cardioplegic solution with deferoxamine on reperfused human myocardium. J Thorac Cardiovasc Surg. 1990 Nov;100(5):708-14. PMID 2232833
- [Background] Menasche P, Pasquier C, Bellucci S, Lorente P, Jaillon P, Piwnica A. Deferoxamine reduces neutrophil-mediated free radical production during cardiopulmonary bypass in man. J Thorac Cardiovasc Surg. 1988 Oct;96(4):582-9. PMID 2845199
- [Background] Menasche P, Antebi H, Alcindor LG, Teiger E, Perez G, Giudicelli Y, Nordmann R, Piwnica A. Iron chelation by deferoxamine inhibits lipid peroxidation during cardiopulmonary bypass in humans. Circulation. 1990 Nov;82(5 Suppl):IV390-6. PMID 2225430
- [Background] Zheng H, Dimayuga C, Hudaihed A, Katz SD. Effect of dexrazoxane on homocysteine-induced endothelial dysfunction in normal subjects. Arterioscler Thromb Vasc Biol. 2002 Jul 1;22(7):E15-8. doi: 10.1161/01.atv.0000023187.25914.5b. PMID 12117747
- [Background] Junjing Z, Yan Z, Baolu Z. Scavenging effects of dexrazoxane on free radicals. J Clin Biochem Nutr. 2010 Nov;47(3):238-45. doi: 10.3164/jcbn.10-64. Epub 2010 Oct 29. PMID 21103033
- [Background] Popelova O, Sterba M, Haskova P, Simunek T, Hroch M, Guncova I, Nachtigal P, Adamcova M, Gersl V, Mazurova Y. Dexrazoxane-afforded protection against chronic anthracycline cardiotoxicity in vivo: effective rescue of cardiomyocytes from apoptotic cell death. Br J Cancer. 2009 Sep 1;101(5):792-802. doi: 10.1038/sj.bjc.6605192. Epub 2009 Jul 21. PMID 19623174
- [Background] Zhou L, Sung RY, Li K, Pong NH, Xiang P, Shen J, Ng PC, Chen Y. Cardioprotective effect of dexrazoxane in a rat model of myocardial infarction: anti-apoptosis and promoting angiogenesis. Int J Cardiol. 2011 Oct 20;152(2):196-201. doi: 10.1016/j.ijcard.2010.07.015. Epub 2010 Aug 6. PMID 20692056
- [Background] Spagnuolo RD, Recalcati S, Tacchini L, Cairo G. Role of hypoxia-inducible factors in the dexrazoxane-mediated protection of cardiomyocytes from doxorubicin-induced toxicity. Br J Pharmacol. 2011 May;163(2):299-312. doi: 10.1111/j.1476-5381.2011.01208.x. PMID 21232037 (Retraction: PMID 32512636 Br J Pharmacol. 2020 Jul;177(13):3123)
- [Background] Hasinoff BB, Schroeder PE, Patel D. The metabolites of the cardioprotective drug dexrazoxane do not protect myocytes from doxorubicin-induced cytotoxicity. Mol Pharmacol. 2003 Sep;64(3):670-8. doi: 10.1124/mol.64.3.670. PMID 12920203
- [Background] Wiseman LR, Spencer CM. Dexrazoxane. A review of its use as a cardioprotective agent in patients receiving anthracycline-based chemotherapy. Drugs. 1998 Sep;56(3):385-403. doi: 10.2165/00003495-199856030-00009. PMID 9777314
- [Background] Brier ME, Gaylor SK, McGovren JP, Glue P, Fang A, Aronoff GR. Pharmacokinetics of dexrazoxane in subjects with impaired kidney function. J Clin Pharmacol. 2011 May;51(5):731-8. doi: 10.1177/0091270010369675. Epub 2010 May 19. PMID 20484616
- [Background] Lipshultz SE, Rifai N, Dalton VM, Levy DE, Silverman LB, Lipsitz SR, Colan SD, Asselin BL, Barr RD, Clavell LA, Hurwitz CA, Moghrabi A, Samson Y, Schorin MA, Gelber RD, Sallan SE. The effect of dexrazoxane on myocardial injury in doxorubicin-treated children with acute lymphoblastic leukemia. N Engl J Med. 2004 Jul 8;351(2):145-53. doi: 10.1056/NEJMoa035153. PMID 15247354
- [Background] Elbl L, Hrstkova H, Tomaskova I, Michalek J. Late anthracycline cardiotoxicity protection by dexrazoxane (ICRF-187) in pediatric patients: echocardiographic follow-up. Support Care Cancer. 2006 Feb;14(2):128-36. doi: 10.1007/s00520-005-0858-8. Epub 2005 Jul 21. PMID 16034614
- [Background] Sanchez-Medina J, Gonzalez-Ramella O, Gallegos-Castorena S. The effect of dexrazoxane for clinical and subclinical cardiotoxicity in children with acute myeloid leukemia. J Pediatr Hematol Oncol. 2010 May;32(4):294-7. doi: 10.1097/MPH.0b013e3181d321b3. PMID 20404753
- [Background] Choi HS, Park ES, Kang HJ, Shin HY, Noh CI, Yun YS, Ahn HS, Choi JY. Dexrazoxane for preventing anthracycline cardiotoxicity in children with solid tumors. J Korean Med Sci. 2010 Sep;25(9):1336-42. doi: 10.3346/jkms.2010.25.9.1336. Epub 2010 Aug 12. PMID 20808678
- [Background] Tebbi CK, London WB, Friedman D, Villaluna D, De Alarcon PA, Constine LS, Mendenhall NP, Sposto R, Chauvenet A, Schwartz CL. Dexrazoxane-associated risk for acute myeloid leukemia/myelodysplastic syndrome and other secondary malignancies in pediatric Hodgkin's disease. J Clin Oncol. 2007 Feb 10;25(5):493-500. doi: 10.1200/JCO.2005.02.3879. PMID 17290056
- [Background] Barry EV, Vrooman LM, Dahlberg SE, Neuberg DS, Asselin BL, Athale UH, Clavell LA, Larsen EC, Moghrabi A, Samson Y, Schorin MA, Cohen HJ, Lipshultz SE, Sallan SE, Silverman LB. Absence of secondary malignant neoplasms in children with high-risk acute lymphoblastic leukemia treated with dexrazoxane. J Clin Oncol. 2008 Mar 1;26(7):1106-11. doi: 10.1200/JCO.2007.12.2481. PMID 18309945
- [Background] Lipshultz SE, Scully RE, Lipsitz SR, Sallan SE, Silverman LB, Miller TL, Barry EV, Asselin BL, Athale U, Clavell LA, Larsen E, Moghrabi A, Samson Y, Michon B, Schorin MA, Cohen HJ, Neuberg DS, Orav EJ, Colan SD. Assessment of dexrazoxane as a cardioprotectant in doxorubicin-treated children with high-risk acute lymphoblastic leukaemia: long-term follow-up of a prospective, randomised, multicentre trial. Lancet Oncol. 2010 Oct;11(10):950-61. doi: 10.1016/S1470-2045(10)70204-7. Epub 2010 Sep 16. PMID 20850381
- [Background] Vrooman LM, Neuberg DS, Stevenson KE, Asselin BL, Athale UH, Clavell L, Cole PD, Kelly KM, Larsen EC, Laverdiere C, Michon B, Schorin M, Schwartz CL, Cohen HJ, Lipshultz SE, Silverman LB, Sallan SE. The low incidence of secondary acute myelogenous leukaemia in children and adolescents treated with dexrazoxane for acute lymphoblastic leukaemia: a report from the Dana-Farber Cancer Institute ALL Consortium. Eur J Cancer. 2011 Jun;47(9):1373-9. doi: 10.1016/j.ejca.2011.03.022. Epub 2011 Apr 20. PMID 21514146
- [Background] Holcenberg JS, Tutsch KD, Earhart RH, Ungerleider RS, Kamen BA, Pratt CB, Gribble TJ, Glaubiger DL. Phase I study of ICRF-187 in pediatric cancer patients and comparison of its pharmacokinetics in children and adults. Cancer Treat Rep. 1986 Jun;70(6):703-9. PMID 3089595
- [Background] Reichardt P, Tabone MD, Mora J, Morland B, Jones RL. Risk-benefit of dexrazoxane for preventing anthracycline-related cardiotoxicity: re-evaluating the European labeling. Future Oncol. 2018 Oct;14(25):2663-2676. doi: 10.2217/fon-2018-0210. Epub 2018 May 11. PMID 29747541
- [Background] Cvetkovic RS, Scott LJ. Dexrazoxane : a review of its use for cardioprotection during anthracycline chemotherapy. Drugs. 2005;65(7):1005-24. doi: 10.2165/00003495-200565070-00008. PMID 15892593
- [Background] Herman, E.H., Hasinoff, B.B., Steiner, R., Lipshultz, S.E. 2014. A review of the preclinical development of dexrazoxane. Prog Ped Card. 36: 33-38
- [Background] Hoffman TM, Wernovsky G, Atz AM, Kulik TJ, Nelson DP, Chang AC, Bailey JM, Akbary A, Kocsis JF, Kaczmarek R, Spray TL, Wessel DL. Efficacy and safety of milrinone in preventing low cardiac output syndrome in infants and children after corrective surgery for congenital heart disease. Circulation. 2003 Feb 25;107(7):996-1002. doi: 10.1161/01.cir.0000051365.81920.28. PMID 12600913
- [Background] Sznycer-Taub N, Mackie S, Peng YW, Donohue J, Yu S, Aiyagari R, Charpie J. Myocardial Oxidative Stress in Infants Undergoing Cardiac Surgery. Pediatr Cardiol. 2016 Apr;37(4):746-50. doi: 10.1007/s00246-016-1345-3. Epub 2016 Feb 3. PMID 26843460
- [Background] Butts RJ, Scheurer MA, Zyblewski SC, Wahlquist AE, Nietert PJ, Bradley SM, Atz AM, Graham EM. A composite outcome for neonatal cardiac surgery research. J Thorac Cardiovasc Surg. 2014 Jan;147(1):428-33. doi: 10.1016/j.jtcvs.2013.03.013. Epub 2013 Apr 12. PMID 23587468
- [Background] Su XW, Undar A. Brain protection during pediatric cardiopulmonary bypass. Artif Organs. 2010 Apr;34(4):E91-102. doi: 10.1111/j.1525-1594.2009.00963.x. PMID 20420605
- [Background] Vidrio H, Carrasco OF, Rodriguez R. Antivasoconstrictor effect of the neuroprotective agent dexrazoxane in rat aorta. Life Sci. 2006 Dec 14;80(2):98-104. doi: 10.1016/j.lfs.2006.08.025. Epub 2006 Aug 25. PMID 17007888
- [Background] Florio P, Abella RF, de la Torre T, Giamberti A, Luisi S, Butera G, Cazzaniga A, Frigiola A, Petraglia F, Gazzolo D. Perioperative activin A concentrations as a predictive marker of neurologic abnormalities in children after open heart surgery. Clin Chem. 2007 May;53(5):982-5. doi: 10.1373/clinchem.2006.077149. Epub 2007 Mar 15. PMID 17363421
- [Background] Fiser DH. Assessing the outcome of pediatric intensive care. J Pediatr. 1992 Jul;121(1):68-74. doi: 10.1016/s0022-3476(05)82544-2. PMID 1625096
- [Background] Mou SS, Giroir BP, Molitor-Kirsch EA, Leonard SR, Nikaidoh H, Nizzi F, Town DA, Roy LC, Scott W, Stromberg D. Fresh whole blood versus reconstituted blood for pump priming in heart surgery in infants. N Engl J Med. 2004 Oct 14;351(16):1635-44. doi: 10.1056/NEJMoa041065. PMID 15483282